CLINICAL TRIAL: NCT02525744
Title: Pharmacokinetics, Glucodynamics, Safety, and Tolerability of a Novel LY900014 Formulation
Brief Title: A Study of a New LY900014 Formulation in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 15989; I8B-FW-ITRE (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY900014 7.5 Units (U) (Experimental): Single dose of 7.5 U LY900014 administered subcutaneously (SC) in one to two of five periods.
  Interventions: Drug: LY900014
- Insulin Lispro (Active Comparator): Reference formulation. Single dose of Insulin Lispro administered SC in one to two of five periods.
  Interventions: Drug: Insulin Lispro (Humalog)
- LY900014 15 U (Experimental): Single dose of 15 U LY900014 administered subcutaneously (SC) in one to two of five periods.
  Interventions: Drug: LY900014
- LY900014 30 U (Experimental): Single dose of 30 U LY900014 administered subcutaneously (SC) in one to two of five periods.
  Interventions: Drug: LY900014

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 15 U; LY900014 30 U; LY900014 7.5 Units (U)
Drug: Insulin Lispro (Humalog) — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro

SUMMARY:
This study evaluates a new formulation of LY900014, a drug that lowers blood sugar. It is administered by injection under the skin of the abdomen. The study will be conducted in healthy people to investigate how quickly and how much LY900014 is absorbed and the effect of different doses of LY900014 on blood sugar levels. Side effects and tolerability will be documented. The study will last for about 8 to 9 weeks for each participant, including screening and follow up. Screening is required within 28 days prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female (not pregnant and agreeable to take birth control measures until one month after study completion)
* Have a body mass index (BMI) of 18.5 to 30 kilogram per square meter (kg/m^2), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Are nonsmokers, have not smoked for at least 2 months prior to entering the study, and agree not to smoke (cigars, cigarettes, or pipes) or use smokeless tobacco for the duration of the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 CBARC: Participants receive single subcutaneous dose:
  C: 30 U LY900014 B: 15 U LY900014 A: 7.5 Units (U) LY900014 R: 15 U insulin lispro(Reference) C: 30 U LY900014
  with 3 day washout between doses
- Sequence 2 ACRBA: Participants receive single subcutaneous dose:
  A: 7.5 Units (U) LY900014 C: 30 U LY900014 R: 15 U insulin lispro(Reference) B: 15 U LY900014 A: 7.5 Units (U) LY900014
  with 3 day washout between doses
- Sequence 3 BRCAB: Participants receive single subcutaneous dose:
  B: 15 U LY900014 R: 15 U insulin lispro(Reference) C: 30 U LY900014 A: 7.5 Units (U) LY900014 B: 15 U LY900014
  with 3 day washout between doses
- Sequence 4 RABCR: Participants receive single subcutaneous dose:
  R: 15 U insulin lispro(Reference) A: 7.5 Units (U) LY900014 B: 15 U LY900014 C: 30 U LY900014 R: 15 U insulin lispro(Reference)
  with 3 day washout between doses
Period: Period 1
Arm/Group | Sequence 1 CBARC | Sequence 2 ACRBA | Sequence 3 BRCAB | Sequence 4 RABCR
Started | 6 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 5 | 6
Completed | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence 1 CBARC | Sequence 2 ACRBA | Sequence 3 BRCAB | Sequence 4 RABCR
Started | 6 | 6 | 5 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 5 | 6
Completed | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 CBARC | Sequence 2 ACRBA | Sequence 3 BRCAB | Sequence 4 RABCR
Started | 6 | 6 | 5 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 5 | 6
Completed | 6 | 5 | 5 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 CBARC | Sequence 2 ACRBA | Sequence 3 BRCAB | Sequence 4 RABCR
Started | 6 | 5 | 5 | 6
Received at Least 1 Dose of Study Drug | 6 | 5 | 5 | 6
Completed | 5 | 5 | 5 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence 1 CBARC | Sequence 2 ACRBA | Sequence 3 BRCAB | Sequence 4 RABCR
Started | 5 | 5 | 5 | 6
Received at Least 1 Dose of Study Drug | 4 | 5 | 5 | 6
Completed | 4 | 5 | 5 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Overall Study: All participants who received at least 1 dose of study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 23
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m2)] | 25.23 (2.27)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) : Insulin Lispro Area Under the Concentration Curve Zero to Infinity (AUC[0-∞]) )
Time Frame: 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300, 360, and 420 minutes per period.
Population: Participants who received at least 1 dose of study drug and had evaluable PK profile data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomol per hour per L (pmol.h/L)
Units Other Than Participants: PK Profiles
Groups:
- LY900014 7.5 U: Participants receive single subcutaneous dose of 7.5 Units (U) LY900014
- LY900014 15 U: Participants receive single subcutaneous dose of 15 Units (U) LY900014
- LY900014 30 U: Participants receive single subcutaneous dose of 30 U LY900014
- Insulin Lispro 15 U: Participants receive single subcutaneous dose of 15 U insulin lispro (Reference, Humalog)
Arm/Group | LY900014 7.5 U | LY900014 15 U | LY900014 30 U | Insulin Lispro 15 U
Number analyzed (Participants) | 24 | 24 | 24 | 24
Number analyzed (PK Profiles) | 27 | 27 | 28 | 29
picomol per hour per L (pmol.h/L) | 901 (17) | 1890 (19) | 3970 (15) | 1790 (14)

2. Secondary Outcome: Total Amount of Glucose Infused (Gtot) Over the Duration of Clamp
Time Frame: Every 10 minutes for 30 minutes Predose, Postdose: every 2.5 minutes for 30 minutes, then every 5 minutes until 120 minutes, then every 10 minutes until 300 minutes, then every 20 minutes until 480 minutes
Population: Participants who received at least 1 dose of study drug and had evaluable GD profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams (mg)
Units Other Than Participants: Glucodynamic (GD) Profiles
Arm/Group | LY900014 7.5 U | LY900014 15 U | LY900014 30 U | Insulin Lispro 15 U
Number analyzed (Participants) | 24 | 24 | 24 | 24
Number analyzed (Glucodynamic (GD) Profiles) | 24 | 24 | 25 | 27
milligrams (mg) | 42900 (67) | 82200 (41) | 122000 (35) | 70700 (48)

ADVERSE EVENTS:
Groups:
- 15 U Insulin Lispro (Reference,Humalog): Participants received single subcutaneous dose of 15 U insulin lispro (Reference, Humalog)
- LY900014 7.5 U: Participants received single subcutaneous dose of 7.5 U LY900014
- LY900014 15 U: Participants received single subcutaneous dose of 15 U LY900014
- LY900014 30 U: Participants received single subcutaneous dose of 30 U LY900014
Arm/Group | 15 U Insulin Lispro (Reference,Humalog) | LY900014 7.5 U | LY900014 15 U | LY900014 30 U
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 3/23 | 3/22 | 6/22 | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 U Insulin Lispro (Reference,Humalog) (N=23) | LY900014 7.5 U (N=22) | LY900014 15 U (N=22) | LY900014 30 U (N=23)
Catheter site related reaction (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Infusion site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Infusion site pain (General disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Infusion site reaction (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No